CLINICAL TRIAL: NCT00334958
Title: A Double-Blind, Placebo-Controlled, Parallel-Group Study of Rufinamide Given as Adjunctive Therapy in Patients With Refractory Partial Seizures
Brief Title: Rufinamide Given as Adjunctive Therapy in Participants With Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2080-A001-301; 2016-004944-12 (EudraCT Number)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — rufinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): For 12-day Titration Phase and 12 week Maintenance Phase, placebo tablets matching to rufinamide 400 mg oral tablets will be administered according to the same regimen scheme as described for rufinamide. For 12-day Titration Phase, 1 matching placebo tablet will be administered twice daily and increased by 1 tablet every 3 days up to maximum of 4 matching placebo tablets twice daily (placebo tablet matched to rufinamide total daily dose of 3200 mg). For the 12 week maintenance phase, 4 placebo tablets matching to rufinamide maintenance doses of 1600 mg twice daily (3200 mg total daily dose) will be administered. Similar to the dose reduction permitted in the rufinamide group, participants in placebo group will be allowed only during the Titration Phase to have the dose reduced to 3 tablets twice daily.
  Interventions: Drug: Placebo
- Rufinamide (Active Comparator): For the 12-day Titration Phase, rufinamide will be administered orally in doses starting with 400 milligram (mg) twice daily and increased every 3 days in 400 mg twice daily increments up to 1600 mg twice daily (total daily dose 3200 mg). For the 12 week Maintenance Phase, maintenance doses of 1600 mg twice daily (3200 mg total daily dose) will be administered. Participants unable to tolerate the target dose (3200 mg/day) will be allowed only during the Titration Phase to have the dose reduced to 3 tablets twice daily (corresponding to a dose of 2400 mg/day in the rufinamide group).
  Interventions: Drug: Rufinamide

INTERVENTIONS:
Drug: Placebo — For the 12-day Titration Phase, one matching placebo tablet will be administered twice daily and increased by 1 matching placebo tablet every 3 days up to maximum of 4 matching placebo tablets twice daily (placebo tablet matched to rufinamide total daily dose of 3200 mg). For the 12 week maintenance phase, 4 placebo tablets matching to rufinamide maintenance doses of 1600 mg twice daily (3200 mg total daily dose) will be administered. Similar to the dose reduction permitted in the rufinamide group, participants in placebo group will be allowed only during the Titration Phase to have the dose reduced to 3 placebo tablets twice daily.
  Arms: Placebo
Drug: Rufinamide — For the titration phase, Rufinamide will be administered orally in doses starting with 400 mg twice daily and increased every 3 days in 400 mg twice daily increments up to 1600 mg twice daily (total daily dose 3200 mg). For the Maintenance Phase, maintenance doses of 1600 mg twice daily (3200 mg total daily dose) will be administered. Participants unable to tolerate the target dose (3200 mg/day) will be allowed only during the Titration Phase to have the dose reduced to 3 tablets twice daily (corresponding to a dose of 2400 mg/day in the rufinamide group).
  Other Names: E2080; BANZEL
  Arms: Rufinamide

SUMMARY:
To evaluate the effect of rufinamide on total partial seizure frequency in adolescent and adult participants (12 to 80 years, inclusive) with refractory partial onset seizures maintained on a maximum of 3 stable antiepileptic drugs (AEDs).

ELIGIBILITY:
INCLUSION CRITERIA

1. Male and female patients between 12 and 80 years of age, inclusive.
2. Diagnosis of epilepsy with partial-onset seizures with or without secondarily generalized seizures according with the International League Against Epilepsy Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history, electroencephalogram (EEG) and computed tomography/magnetic resonance imaging (CT/MRI) of the brain performed within the last 10 years and consistent with localization-related epilepsy.
3. Non-controlled partial seizures despite having been treated with at least two different antiepileptic drugs (given concurrently or sequentially) for at least two years.
4. Patient willing to participate and written consent signed by patient or legal guardian prior to entering the study or undergoing any study procedures. If the written consent is provided by a legal guardian because the patient is unable to do so, assent of the patient must also be obtained.
5. Reliability and willingness of patients to make themselves available for the study period, and ability to record seizures and report adverse events themselves or have a caregiver who can record seizures and report adverse events.
6. Female patients of non-childbearing potential by reason of surgery, radiation, or menopause (at least one year post onset); or of childbearing potential using two approved methods of contraception (such as an intrauterine device [IUD], implant, oral contraceptive, or barrier method plus spermicide). Use of a low-dose estrogen oral contraceptive ("minipill") alone will not be permitted. Female patients of childbearing potential must have a confirmed negative serum pregnancy test at screening and a negative urine pregnancy test prior to randomization, and agree to continue to use two approved methods of contraception through the follow-up visit (Visit 8) or for 30 days after their final dose of study medication, whichever is longer.
7. At least six seizures during the prospective Baseline Phase (56 days) with no 21-day seizure-free periods. Simple partial seizures without motor signs will not be included in determining this criterion.
8. Current treatment with a maximum of three approved antiepileptic drugs, and no evidence of non-compliance with ongoing AED therapy.
9. Stable dose(s) of the same AED(s) for one month prior to screening.
10. If using a vagal nerve stimulator, it must have been implanted for at least six months prior to randomization. Stimulator parameters may not be changed for at least one month prior to screening or thereafter during the study. Magnet use will be allowed, but must be documented throughout the study. A vagal nerve stimulator will not be counted as an AED for the purpose of inclusion into the trial.

EXCLUSION CRITERIA:

1. Participation in a study involving administration of an investigational compound within one month of Visit 1 (Screening), or within five half-lives of the previous investigational compound, whichever is longer; or any prior exposure to rufinamide.
2. Presence of non-motor simple partial seizures only.
3. Presence of generalized epilepsies or seizures, such as absences, myoclonic epilepsies, Lennox-Gastaut syndrome.
4. History of status epilepticus in the past year or seizure clusters where individual seizures cannot be counted.
5. Evidence of clinically significant disease (cardiac, respiratory, gastrointestinal, hepatic, hematologic or renal disease, etc.) that in the opinion of the Investigator could affect the patient's safety or trial conduct.
6. Clinically significant ECG abnormality.
7. Patients with a diagnosis of major active psychiatric disease will be excluded from the study. However, those patients who are only taking a stable dose of either a selective serotonin reuptake inhibitor (SSRI) antidepressant drug or a serotonin and norepinephrine reuptake inhibitor (SNRI) antidepressant drug for a diagnosed depressive disorder can be included as long as they have been on the SSRI or SNRI for a period of two months or longer before randomization. Other antidepressant medications will not be allowed.
8. Progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
9. Occurrence of psychogenic seizures in the previous year.
10. History of drug abuse and/or positive finding on urinary drug screening, other than prescribed medication
11. History of alcohol abuse in the past two years.
12. History of suicide attempt within the previous 10 years.
13. Multiple drug allergies (dermatological, hematological or organ toxicity) or more than one severe drug reaction(s).
14. Concomitant use of felbamate or use of felbamate within two months prior to Visit 1.
15. Frequent need of rescue benzodiazepines (more than once a month).
16. Patients with a known hypersensitivity to rufinamide, triazole derivatives, or to any excipients used in the formulation.
17. Concomitant use of vigabatrin. Patients who took vigabatrin in the past must be off vigabatrin for at least five months prior to Visit 1 and must not have evidence of a clinically significant abnormality in a visual perimetry test.
18. All Patients with a diagnosis of Congenital Short QT Syndrome. Patients with a family history of Congenital Short QT Syndrome may be excluded on the basis of the Investigator's clinical judgment.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2006-02-13 (Actual); Primary Completion 2009-05-20 (Actual); Study Completion 2009-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (77):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Neurology Clinic PC, Northport, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Epilepsy and Neurology, Phoenix, Arizona
  - University of Arizona, Dept. of Neurology, Tucson, Arizona
  - Clinical Trials, Inc, Little Rock, Arkansas
  - Neuro-Pain Medical Center, Inc., Fresno, California
  - Neurology Center, Oceanside, California
  - California Pacific Epilepsy, San Francisco, California
  - Georgetown University Hospital, Dept. of Neurology, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Bradenton Research Center, Bradenton, Florida
  - University of Florida, Dept. of Neurology, Gainesville, Florida
  - University of Florida, The Neuroscience Institute at Shands, Jacksonville, Florida
  - Pediatric Neurologists of Palm Beach, Loxahatchee Groves, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Pediatric Neurology - PA, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - University of Southern Florida, Dept. of Neurology, Tampa, Florida
  - Child Neurology Associates, PC, Atlanta, Georgia
  - Medical College of Georgia, Dept. of Neurology, Augusta, Georgia
  - Medical Associates of North Georgia, Canton, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Children's Memorial Hospital, Northwest University, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Children's Hospital, Park Ridge, Illinois
  - Southern Illinois University Neurology and Pharmacology, Springfield, Illinois
  - Mcfarland Clinic, Ames, Iowa
  - Via Christi Comprehensive Epilepsy Center, Wichita, Kansas
  - University of Kentucky, Dept. of Neurology, Lexington, Kentucky
  - John Hopkins Hospital, Dept. of Neurology, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Boston University Medical Center, Dept. of Neurology, Boston, Massachusetts
  - University of Massachusetts, Neurology Associates, Hopedale, Massachusetts
  - University of Minnesota, Dept. of Neurology, Minneapolis, Minnesota
  - Minnesota Epilepsy Group, PC, Saint Paul, Minnesota
  - Ronald Schwartz, M.D., Hattiesburg, Mississippi
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Saint John's Medical Research, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Dartmouth Medical School Neuroscience Center, Lebanon, New Hampshire
  - Five Towns Neuroscience Research, Lawrence, New York
  - New York University Medical Centre, Comprehensive Epilepsy Center, New York, New York
  - Weill Cornell Medical Center, Comprehensive Epilepsy Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Dept. of Neurology, Chapel Hill, North Carolina
  - Duke Health Center at Morreene Road, Durham, North Carolina
  - Cleveland Clinic Foundation, Dept. of Neurology, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of Ohio at Toledo, Dept. of Neurology, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Blair Medical Associates, Inc., Altoona, Pennsylvania
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Dept. of Neurology, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh - Dept of Pediatrics, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Mid-South Physicians Group, PLLC, Germantown, Tennessee
  - University of Tennessee Health Sciences Center, Dept. of Neurology, Memphis, Tennessee
  - UT Medical Group, Memphis, Tennessee
  - Access Clinical Trials, Inc, Nashville, Tennessee
  - Neurological Clinic of Texas, PA, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Tech University Health Sciences Center, Dept. of Neuropsychiatry, El Paso, Texas
  - University of Texas - Dept of Neurology, Houston, Texas
  - Baylor Medical Center of Irving, Irving, Texas
  - Epilepsy and Neurodevelopment, Inc., West Jordan, Utah
  - University of Vermont, College of Medicine, Clinical Neurophysiology Lab, Burlington, Vermont
  - Fletcher Allen Healthcare, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Harborview Medical Center, Regional Epilepsy Center, Seattle, Washington
  - University of Wisconsin, Dept. of Neurology, Madison, Wisconsin

REFERENCES:
- [Derived] Panebianco M, Prabhakar H, Marson AG. Rufinamide add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2020 Nov 8;11(11):CD011772. doi: 10.1002/14651858.CD011772.pub3. PMID 33179247

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened at 75 centers (69 in the United States and 6 in Canada). Participants were enrolled at 65 centers (61 in the United States and 4 in Canada).
Groups:
- Rufinamide: For the 12-day Titration Phase, rufinamide were administered orally in doses starting with 400 mg twice daily and increased every 3 days in 400 mg twice daily increments up to 1600 mg twice daily (total daily dose 3200 mg). For the 12 week Maintenance Phase, maintenance doses of 1600 mg twice daily (3200 mg total daily dose) were administered. Participants unable to tolerate the target dose (3200 mg/day) were allowed only during the Titration Phase to have the dose reduced to 3 tablets twice daily (corresponding to a dose of 2400 mg/day in the rufinamide group).
- Placebo: For 12-day Titration Phase and 12 week Maintenance Phase, placebo tablets matching to rufinamide 400 mg oral tablets were administered according to the same regimen scheme as described for rufinamide. For 12-day Titration Phase, 1 matching placebo tablet were administered twice daily and increased by 1 tablet every 3 days up to maximum of 4 matching placebo tablets twice daily (placebo tablet matched to rufinamide total daily dose of 3200 mg). For the 12 week maintenance phase, 4 placebo tablets matching to rufinamide maintenance doses of 1600 mg twice daily (3200 mg total daily dose) were administered. Similar to the dose reduction permitted in the rufinamide group, participants in placebo group were allowed only during the Titration Phase to have the dose reduced to 3 tablets twice daily.
Period: Overall Study
Arm/Group | Rufinamide | Placebo
Started | 176 | 180 (1 participant withdrawn prior to study drug dosing due to not obtaining labs)
Completed | 139 | 156
Not Completed | 37 | 24
Not completed — Medication Noncompliance | 0 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Request of the investigator or sponsor | 0 | 1
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Adverse Event | 27 | 12
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rufinamide | Placebo | Total
Number analyzed (Participants) | 176 | 180 | 356
Age, Customized [Number; unit: participants] — Safety population
  participants
    12 to < 18 years | 15 | 21 | 36
    18 to <65 years | 155 | 153 | 308
    >=65 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population: All randomized participants who received at least 1 dose of study medication.
  Participants
    Female | 92 | 97 | 189
    Male | 84 | 83 | 167
Race/Ethnicity, Customized [Number; unit: participants] — Race (Safety population)
  participants
    Black | 14 | 19 | 33
    White | 145 | 140 | 285
    Hispanic | 13 | 14 | 27
    Native American | 0 | 2 | 2
    Asian/Pacific Islander | 4 | 2 | 6
    Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Total Partial Seizure Frequency Per 28 Days During Maintenance Phase Relative to the Baseline Phase
Description: Seizure data was collected via patient diary, which was used to record daily seizure count and type. Intent-to-treat (ITT) population: All randomized participants who had baseline Patient Seizure Diary data and had at least completed the titration period.
Time Frame: Baseline, Days 13 to 96
Population: Intent-to-treat (ITT) population: All randomized participants who had baseline Patient Seizure Diary data and had at least completed the titration period.
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 160 | 175
Percentage change | -23.25 [-100.0 to 725.6] | -9.80 [-100.0 to 864.3]

2. Secondary Outcome: Percentage of Participants With 50% or Greater Reduction in Total Partial Seizure Frequency Per 28 Days During the Maintenance Phase Relative to the Baseline Phase
Description: Seizure data was collected via patient diary, which was used to record daily seizure count and type.
Time Frame: Baseline, Days 13 to 96
Population: ITT population: All randomized participants who had baseline Patient Seizure Diary data and had at least completed the titration period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 160 | 175
Percentage of Participants | 32.5 | 14.3

3. Secondary Outcome: Log10 Transformed Total Partial Seizure Frequency Per 28 Days During the Baseline Phase and Maintenance Phase
Description: Total partial seizure frequencies per 28 days during the double-blind Maintenance and Baseline Phases were transformed using logarithms to the base 10 (log10), because it was expected from previous studies that the results would not be normally distributed.
Time Frame: Days 13 to 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Seizures per 28-days (log-transformed)
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 160 | 175
Seizures per 28-days (log-transformed) | 0.98 (0.675) | 1.13 (0.520)

4. Secondary Outcome: Reduction From Baseline in Total Partial Seizure Frequency Rate (RRATIO) During Maintenance Phase
Description: RRATIO= 100*(T-B)/(T+B) where T= total seizure frequency per 28 days during the Maintenance Phase, and B=total seizure frequency per 28 days during the Baseline Phase.
Time Frame: Baseline, Days 13 to 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: RRATIO
Arm/Group | Rufinamide | Placebo
Number analyzed (Participants) | 160 | 175
RRATIO | -18.76 (37.841) | -6.90 (24.869)

ADVERSE EVENTS:
Time Frame: All AEs were collected throughout the study from the time of consent to follow-up visit or 30 days after study drug discontinuation, whichever was longer (up to approximately 3 years and 3 months)
Description: Serious adverse events (SAEs), regardless of causality assessment, were collected through the follow-up visit or 30 days after study drug discontinuation, whichever was longer.
Arm/Group | Rufinamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/180
Serious Adverse Events (participants affected / at risk) | 6/176 | 7/180
Other Adverse Events (participants affected / at risk) | 101/176 | 66/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (N=176) | Placebo (N=180)
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Complex partial seizures (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 2 | 2
Coordination abnormal (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (N=176) | Placebo (N=180)
Diplopia (Eye disorders) | 14 | 2
Nausea (Gastrointestinal disorders) | 22 | 9
Vomiting (Gastrointestinal disorders) | 13 | 9
Fatigue (General disorders) | 27 | 18
Upper respiratory tract infection (Infections and infestations) | 6 | 15
Contusion (Injury, poisoning and procedural complications) | 9 | 5
Dizziness (Nervous system disorders) | 47 | 15
Headache (Nervous system disorders) | 29 | 23
Somnolence (Nervous system disorders) | 22 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No